CLINICAL TRIAL: NCT07239947
Title: A Randomized, Blinded, Placebo-controlled, Single- and Multiple-ascending Dose Study to Evaluate Safety, Tolerability, Pharmacokinetics, Immunogenicity, Pharmacodynamics and Clinical Activity of BBT001 in HVs and AD Patient
Brief Title: A Study of BBT001 in Healthy Volunteers (HVs) and in Adult Patients With Moderate to Severe Atopic Dermatitis (AD)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bambusa Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: BBT001-002
Record Dates: First submitted 2025-09-28; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A -BBT001(Single Ascending Dose) (Experimental): A single dose of BBT001 will be administered in healthy volunteers
  Interventions: Drug: BBT001
- Part A- Placebo(Single Ascending Dose) (Experimental): A single dose of Placebo will be administered in healthy volunteers
  Interventions: Drug: Placebo
- Part B- BBT001(Multiple Ascending Dose) (Experimental): Seven repeat doses of BBT001 will be administered in patients with moderate to severe atopic dermatitis
  Interventions: Drug: BBT001
- Part B -Placebo (Multiple Ascending Dose)) (Experimental): Seven repeat doses of Placebo will be administered in patients with moderate to severe atopic dermatitis
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BBT001 — BBT001 will be administered
  Arms: Part A -BBT001(Single Ascending Dose); Part B- BBT001(Multiple Ascending Dose)
Drug: Placebo — Placebo will be administered
  Arms: Part A- Placebo(Single Ascending Dose); Part B -Placebo (Multiple Ascending Dose))

SUMMARY:
This is a Phase 1, randomized, blinded, placebo controlled, single ascending dose (SAD) study of BBT001 in healthy volunteers (HVs) and adult patients with moderate to severe Atopic Dermatitis (AD).

DETAILED DESCRIPTION:
The study consists of two parts:

Part A (single dose in HVs in sequential ascending dose cohorts, SAD in HVs part) Part B (seven repeated doses in patients with moderate to severe AD, multiple ascending Dose in patients part)

ELIGIBILITY:
Key Inclusion Criteria ( Part A and B):

1. Age of 18-65 years.
2. Body mass index between 18-28 kg/m², capped at 120 kg.
3. Negative pregnancy tests for women of childbearing potential.
4. Willingness to refrain from alcohol consumption for 24 hours prior to each study visit.
5. Non-smokers, healthy current smokers (≤5 cigarettes/day), or ex-smokers.
6. Adequate contraception use (for men and women of childbearing potential).
7. No clinically significant abnormalities or history of relevant diseases.

Key Inclusion Criteria (Part B only):

1. Must have dermatologist-confirmed chronic atopic dermatitis (≥12 months). Inadequate response to topical treatments or where they are medically inadvisable.
2. Moderate to severe atopic dermatitis
3. Validated investigator's global assessment for atopic dermatitis (vIGA-ADTM) score ≥3
4. Atopic lesions cover ≥10% of body surface area (BSA)
5. Average peak pruritus numeric rating scale (PP-NRS) score ≥4 in the 7 days before randomization.
6. Eczema Area and Severity Index (EASI) score ≥16 at screening and randomization visits.

Key Exclusion Criteria for (Part A&B)

1. Significant health issues, such as: diabetes, positive tests for human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B surface antigen (HBsAg), immunodeficiencies, autoimmune diseases, or cancer, history of conditions predisposing to infections.
2. History of major metabolic, dermatological, liver, kidney, hematological, or other significant disorders.
3. Clinically relevant abnormal lab results, including low blood counts, liver issues, or abnormal kidney function.
4. Positive drug/alcohol tests or abnormal vital signs at screening or Day -1.
5. Abnormal Electrocardiogram (ECG) findings
6. History of drug/alcohol abuse in the past 2 years.
7. Donated >500mL blood within 2 months of screening.
8. History of severe allergic reactions or hypersensitivity.

Key Exclusion Criteria for (Part B only)

1. Skin diseases other than atopic dermatitis, significant tattoos, or scarring.
2. Receipt of immunoglobulin or blood products within 30 days.
3. Atopic dermatitis with ocular symptoms or chronic ocular steroid use.
4. Chronic pruritus from conditions other than atopic dermatitis.
5. Acute/treated infections or chronic skin infections.
6. Current use of sedating antihistamines or corticosteroids.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2025-08-09 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-03-26 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events following single and multiple administration of BBT001 | Part A- Up to Day 141; Part B - Up to Day 169 post first dose administration
  Incidence, relatedness, and severity of adverse events graded per NCI CTCAE v5.0.
Number of participants with change in vital sign measurements following treatment administration. | Part A- Up to Day 141; Part B-Up to Day 169 post first dose administration
  Blood pressure and heart rate will be assessed.
Number of participants with change in serum blood parameters. | Part A- Up to Day 141; Part B - Up to Day 169 post first dose administration
  Laboratory assessments include hematology, blood chemistry and coagulation test
Number of participants with change in physical examination following treatment administration. | Part A- Up to Day 141; Part B - Up to Day 169 post first dose administration
  Physical examination will be assessed.
Number of participants with change in 12-lead electrocardiogram (ECG) results measurements following treatment administration. | Part A- Up to Day 141; Part B - Up to Day 169 post first dose administration
  12-lead ECG will be tested at individual sites using sites' equipment and will be assessed.

SECONDARY OUTCOMES:
Pharmacokinetics parameters- maximum observed Concentration (Cmax) | At specified timepoints pre-dose and up to 169 days post first dose administration.
  Maximum observed concentration of the study drug in serum will be analyzed for all subjects.
Pharmacokinetics parameters- Time for maximum observed Concentration (Tmax) | At specified timepoints pre-dose and up to 169 days post first dose administration
  Serum PK Tmax will be analyzed for all subjects
Pharmacokinetics parameters- Area under the curve (AUC) | At specified timepoints pre-dose and up to 169 days post first dose administration
  Area under the curve of the study drug in serum will be analyzed for all subjects
Pharmacokinetics parameters- Volume of distribution (Vz) | At specified timepoints pre-dose and up to 169 days post first dose administration
  Volume of distribution of the study drug in serum will be analyzed for all subjects
Pharmacokinetics parameters- Total clearance (CL) | At specified timepoints pre-dose and up to 169 days post first dose administration
  Total clearance of the study drug in serum will be analyzed for all subjects
Pharmacokinetics parameters- - Elimination Half-life (t1/2). | At specified timepoints pre-dose and up to 169 days post first dose administration
  Elimination half-life of the study drug in serum will be analyzed for all subjects
The immunogenicity of BBT001 is measured as the number and percentage of subjects who develop Anti-Drug Antibodies (ADA). | At specified timepoints pre-dose and up to 169 days post first dose administration
  Serum Anti-Drug Antibodies will be analyzed for all subjects

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Ji, Study Director — Bambusa (Beijing) Therapeutics Co., Ltd.
Locations (10):
- China (10):
  - The Second Hospital of Anhui Medical Univesity, Hefei, Anhui
  - The Second Affiliated Hospital of Wannan Medical College, Wuhu, Anhui
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Dermatology Hospital of Southern Medical University, Guangzhou, Guangdong
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Wuxi Second People's Hospital, Wuxi, Jiangsu
  - Jiangsu University Affiliated Hospital, Zhenjiang, Jiangsu
  - Jiangxi Provincial Dermatology Hospital, Nanchang, Jiangxi
  - Shandong Provincial Hospital for Skin Diseases, Jinan, Shandong
  - Shanghai Dermatology Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No